CLINICAL TRIAL: NCT06173583
Title: ARISCAT and LAS VEGUS Risk Scores for Predicting Postoperative Pulmonary Complications After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Khalid Siddiqui, Associate Professor, Aga Khan University
Other Study IDs: 2020-1743-8434
Record Dates: First submitted 2023-12-08; First posted 2023-12-15 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Complication; Postoperative Complications; Postoperative Pulmonary Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult In-patient Cardiac surgery: Adult patients undergoing elective open-heart surgery
  Interventions: Diagnostic Test: Detection/screening

INTERVENTIONS:
Diagnostic Test: Detection/screening — Using ARISCAT and LAS VEGUS risk scores for predicting PPCs

SUMMARY:
The goal of this observational study is to compare the, ARISCAT and LAS VEGUS scales, for predicting postoperative pulmonary complications in patients undergoing cardiac surgery. The study aims to compare the diagnostic accuracies of the two risk prediction scores in predicting postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective heart surgery

Exclusion Criteria:

* Refusal to consent
* Patients undergoing emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either gender, aged between 18-65 years, undergoing elective heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of ARISCAT and LAS VEGAS Scoring systems | Day 1-5
  Diagnostic Accuracy to judge the Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) and Local Assessment of Ventilatory Management During General Anaesthesia for Surgery (LAS VEGAS) Scoring systems to predict Postoperative Pulmonary Complications (PPC) after Cardiac surgery. Scores, ARISCAT ≥ 27 and LAS VEGAS ≥ 8 were determined for PPCs.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan